CLINICAL TRIAL: NCT02139943
Title: A Randomized Phase 2, Double-blind, Placebo-controlled, Treat-to-Target, Parallel-group, 3-arm, Multicenter Study to Assess the Efficacy and Safety of Canagliflozin as Add-on Therapy to Insulin in the Treatment of Subjects With Type 1 Diabetes Mellitus
Brief Title: A Study of Effects of Canagliflozin as Add-on Therapy to Insulin in the Treatment of Participants With Type 1 Diabetes Mellitus (T1DM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR104173; 2013-005078-24 (EudraCT Number); 28431754DIA2004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Results first posted 2016-07-18 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Canagliflozin; Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Canagliflozin 100 mg (Experimental): Each participant will receive 100 mg of canagliflozin once daily for 18 weeks.
  Interventions: Drug: Canagliflozin 100 mg
- Canagliflozin 300 mg (Experimental): Each participant will receive 300 mg of canagliflozin once daily for 18 weeks.
  Interventions: Drug: Canagliflozin 300 mg
- Placebo (Placebo Comparator): Each participant will receive matching placebo once daily for 18 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin 100 mg — Canagliflozin capsule of 100 mg dose will be taken orally, before the first meal of the day.
  Arms: Canagliflozin 100 mg
Drug: Canagliflozin 300 mg — Canagliflozin capsule of 300 mg dose will be taken orally, before the first meal of the day.
  Arms: Canagliflozin 300 mg
Drug: Placebo — Matching placebo capsule will be taken orally, before the first meal of the day.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effects of administration of canagliflozin 100 mg and 300 mg, compared with placebo as an addition to insulin therapy for the treatment of Type 1 Diabetes Mellitus (T1DM).

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), double-blind (neither physician nor participant knows the identity of the assigned treatment), placebo-controlled (an inactive substance that is compared with a medication to test whether the medication has a real effect) parallel-group, multicenter study of canagliflozin as an addition to insulin therapy for participants with type 1 diabetes mellitus and inadequate glycemic control.

Approximately 330 participants will be randomly assigned in a 1:1:1 ratio to either canagliflozin 100 mg, canagliflozin 300 mg, or placebo groups. About 90 participants (30 per treatment group) will be selected for a substudy with a purpose of a continuous glucose monitoring (CGM) assessment for 7 days at baseline and 7 days at the end of treatment.

The total duration of the participation will be about 22 weeks, during which participants will need to return to investigational sites for approximately 9 visits. During the study participants will receive advice on treatment of hypoglycemia and diabetic ketoacidosis (DKA), as well as on compliance with diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Must have type 1 diabetes mellitus (T1DM) for at least 1 year
* Must have have inadequate glycemic control (as defined by glycosylated hemoglobin level of >= 7.0% to <= 9.0%) on basal plus bolus insulin at screening
* Must have body mass index 21 to 35 kg/m2 inclusive
* Must be on a total daily dose of insulin >= 0.6 IU/kg at screening
* Must be on a stable insulin regimen for at least 8 weeks prior to screening

Exclusion Criteria:

* History of T2DM, pancreas or β-cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy
* Severe hypoglycemia (defined as an event required assistance from another person, or which resulted in seizure or loss of consciousness) within 6 months prior to study start
* Diabetic ketoacidosis within 6 months prior to study start
* History of hereditary glucose-galactose malabsorption or primary renal glycosuria
* An ongoing, inadequately controlled thyroid disorder

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (53):
- United States (46):
  - Little Rock, Arkansas
  - Concord, California
  - La Jolla, California
  - Los Angeles, California
  - Los Gatos, California
  - Northridge, California
  - Orange, California
  - San Francisco, California
  - Temecula, California
  - Tustin, California
  - Ventura, California
  - Walnut Creek, California
  - Denver, Colorado
  - Miami, Florida
  - Palm Harbor, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Council Bluffs, Iowa
  - Des Moines, Iowa
  - Baton Rouge, Louisiana
  - Rockville, Maryland
  - Billings, Montana
  - Omaha, Nebraska
  - El Paso, Nevada
  - Las Vegas, Nevada
  - Nashua, New Hampshire
  - Billings, New York
  - Smithtown, New York
  - Morehead City, North Carolina
  - Columbus, Ohio
  - Mentor, Ohio
  - Philadelphia, Pennsylvania
  - Greer, South Carolina
  - Bloomington, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Schertz, Texas
  - Tomball, Texas
  - Ogden, Utah
  - Salt Lake City, Utah
  - Spokane, Washington
  - Milwaukee, Wisconsin
- Canada (7):
  - Calgary, Alberta
  - London, Ontario
  - Oakville, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
  - Laval, Quebec
  - Sainte-Foy, Quebec

REFERENCES:
- [Derived] Rodbard HW, Peters AL, Slee A, Cao A, Traina SB, Alba M. The Effect of Canagliflozin, a Sodium Glucose Cotransporter 2 Inhibitor, on Glycemic End Points Assessed by Continuous Glucose Monitoring and Patient-Reported Outcomes Among People With Type 1 Diabetes. Diabetes Care. 2017 Feb;40(2):171-180. doi: 10.2337/dc16-1353. Epub 2016 Nov 29. PMID 27899497
- [Derived] Peters AL, Henry RR, Thakkar P, Tong C, Alba M. Diabetic Ketoacidosis With Canagliflozin, a Sodium-Glucose Cotransporter 2 Inhibitor, in Patients With Type 1 Diabetes. Diabetes Care. 2016 Apr;39(4):532-8. doi: 10.2337/dc15-1995. PMID 26989182
- [Derived] Henry RR, Thakkar P, Tong C, Polidori D, Alba M. Efficacy and Safety of Canagliflozin, a Sodium-Glucose Cotransporter 2 Inhibitor, as Add-on to Insulin in Patients With Type 1 Diabetes. Diabetes Care. 2015 Dec;38(12):2258-65. doi: 10.2337/dc15-1730. Epub 2015 Oct 20. PMID 26486192

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 614 participants were screened and 352 subjects (57.3%) were randomized to study drug. One subject randomized to placebo did not take any study drug and withdrew consent on the day of randomization.
Groups:
- Placebo: Participants received canagliflozin matching placebo capsules once daily for 18 weeks.
- Canagliflozin 100 Milligram (mg): Participants received 100 mg of canagliflozin capsules once daily for 18 weeks.
- Canagliflozin 300 mg: Participants received 300 mg of canagliflozin capsules once daily for 18 weeks.
Period: Overall Study
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Started | 117 | 117 | 117
Completed | 107 | 111 | 110
Not Completed | 10 | 6 | 7
Not completed — Adverse Event | 0 | 1 | 2
Not completed — Lost to Follow-up | 3 | 2 | 2
Not completed — Withdrawal by Subject | 4 | 3 | 0
Not completed — Other | 0 | 0 | 1
Not completed — Participant wishes to discontinue | 2 | 0 | 0
Not completed — Participant in Poor Compliance | 1 | 0 | 1
Not completed — eGFR Withdrawal Criteria | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat analysis set included all randomized participants who took at least 1 dose of double-blind study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg | Total
Number analyzed (Participants) | 117 | 117 | 117 | 351
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 117 | 115 | 115 | 347
  >=65 years | 0 | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (11.9) | 42 (11.6) | 42.8 (10.96) | 42.3 (11.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 48 | 52 | 154
  Male | 63 | 69 | 65 | 197
Region Enroll [Number; unit: participants]
  Canada | 24 | 19 | 20 | 63
  United Stats | 93 | 98 | 97 | 288

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hemoglobin A1c (HbA1c) Reduction Greater Than or Equal to (>=) 0.4 Percent (%) and no Increase in Body Weight
Description: Clinical response at Weeks 18 was assessed by the percentage of participants with Hemoglobin A1c (HbA1c) reduction greater than or equal to 0.4 % and had no increase in body weight.
Time Frame: Week 18
Population: Modified intent-to-treat analysis set included all randomized participants who took at least 1 dose of double-blind study drug. 'N (Number of Participants Analyzed)' signifies participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Number analyzed (Participants) | 110 | 111 | 111
percentage of participants
  Yes | 14.5 | 36.9 | 41.4
  No | 85.5 | 63.1 | 58.6

2. Primary Outcome: Percentage of Participants With Adverse Events
Time Frame: Up to 22 Weeks
Population: Safety Analysis Set included all randomized participants who took at least 1 dose of double-blind study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Number analyzed (Participants) | 117 | 117 | 117
percentage of participants | 54.7 | 55.6 | 67.5

ADVERSE EVENTS:
Time Frame: Up to 22 Weeks
Arm/Group | Placebo | Canagliflozin 100 Milligram (mg) | Canagliflozin 300 mg
Serious Adverse Events (participants affected / at risk) | 0/117 | 9/117 | 8/117
Other Adverse Events (participants affected / at risk) | 32/117 | 36/117 | 43/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=117) | Canagliflozin 100 Milligram (mg) (N=117) | Canagliflozin 300 mg (N=117)
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 5 | 7
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=117) | Canagliflozin 100 Milligram (mg) (N=117) | Canagliflozin 300 mg (N=117)
Nausea (Gastrointestinal disorders) | 3 | 4 | 6
Nasopharyngitis (Infections and infestations) | 10 | 9 | 6
Sinusitis (Infections and infestations) | 6 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 11 | 10 | 10
Urinary tract infection (Infections and infestations) | 2 | 5 | 6
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 2 | 8
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 7
Pollakiuria (Renal and urinary disorders) | 3 | 5 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.